CLINICAL TRIAL: NCT02729142
Title: Longitudinal Monitoring of Bone Microarchitecture by High Resolution Peripheral Quantitative Computed Tomography of (HR-pQCT) in the Transplant Patient
Brief Title: Bone Microarchitecture in the Transplant Patient
Acronym: TRANSOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL14_0223; 2015-A00510-49 (Other: IDRCB)
Record Dates: First submitted 2016-03-25; First posted 2016-04-06 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2020-11

CONDITIONS: Organ Transplant
Keywords: HRpQCT; transplant; bone microarchitecture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tibial cortical density evaluation (Experimental)
  Interventions: Procedure: Tibial cortical density evaluation

INTERVENTIONS:
Procedure: Tibial cortical density evaluation — Bone evaluation in transplant patients will be performed by HR-pQCT at baseline (either within 6 months before surgery or within 15 days following surgery) and 6 months post-intervention in order to assess its evolution.

SUMMARY:
The optimal management of calcium and phosphate metabolism regulation in chronic kidney disease (CKD) is important in preventing fracture risk and vascular calcification and thus morbidity and mortality, global and vascular.

Kidney transplant in a CKD context, usually with a pre-existing underlying renal osteodystrophy, malnutrition, chronic inflammation, hypogonadism and immunosuppression protocols still often made up of high-dose corticosteroid therapy, are all theoretical factors of post-transplantation bone disease. For other solid organ transplants, even though there is generally no underlying renal osteodystrophy before the transplant, the proportion of osteoporotic patients at the time of transplant is substantial. The bone risk in the immediate post-transplant period is notable.

Patients' follow-up is based on biological, radiological and histological tools. Bone densitometry (DXA) is used to measure bone mass. However, recent international recommendations do not consider DXA as a valid tool to assess bone health in CKD patients. Moreover, it is less informative than peripheral quantitative tomography resolution (HR-pQCT). This latest technique, available in Lyon and Saint-Etienne, is more precise, allowing a three-dimensional study of the trabecular microarchitecture and compartmental volumetric bone density (total, cortical, trabecular), while similar to DXA in terms of radiation (less than 5 μSv). The prevention of cardiovascular risk factors is also part of the daily care of patients with a regular cardiac monitoring (heart ultrasound) and vascular (blood pressure, Doppler of the supra-aortic trunks).

TRANSOS study aims to evaluate in a prospective cohort (longitudinal follow-up of 6 months), the bone status in patients receiving solid organ transplantation in the University Hospitals of Lyon and Saint-Etienne, using DXA and HR-pQCT (at baseline and month 6), in combination with classical biological and cardiovascular monitoring. Transplantation is an important activity in these two hospitals and this protocol provides the same bone follow-up for all solid organ transplants, with a reliable, efficient, non-invasive and low-dose radiation tool.

The primary objective of TRANSOS study is to evaluate changes in tibial cortical density between the baseline and the 6th month post-transplant measured by HR-pQCT.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 10 year-old
* Patient receiving a first solid organ transplant within involved hospitals (Lyon, Saint Etienne): kidney, heart, kidney-pancreas, lung
* Informed consent signed by the patients or their parents (minors)

Exclusion Criteria:

* No health cover
* Ongoing pregnancy

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Tibial cortical density measured by HR-pQCT | at 6 months

SECONDARY OUTCOMES:
trabecular bone area measured by HR-pQCT | at 6 months
total bone area measured by HR-pQCT | at 6 months
trabecular number measured by HR-pQCT | at 6 months
trabecular thickness measured by HR-pQCT | at 6 months
trabecular separation measured by HR-pQCT | at 6 months
cortical perimeter measured by HR-pQCT | at 6 months
Evaluation of bone markers by measuring calcium | at 6 months
Evaluation of bone markers by measuring phosphate | at 6 months
Evaluation of bone markers by measuring alkaline reserve | at 6 months
Evaluation of bone markers by measuring PTH | at 6 months
Evaluation of bone markers by measuring 25OHD3 | at 6 months
Evaluation of bone markers by measuring 1-25 OHD3 | at 6 months
Evaluation of bone markers by measuring FGF23 | at 6 months
Evaluation of bone markers by measuring CTX | at 6 months
Evaluation of bone markers by measuring total alkaline phosphatase | at 6 months
Evaluation of bone markers by measuring bone alkaline phosphatase | at 6 months
Evaluation of bone markers by measuring osteocalcin | at 6 months
Bone mineral density assessed by DXA | at 6 months
Fractures onset assessed by DXA | at 6 months
Cardiovascular events (death from cardiovascular cause, heart attack, stroke) | at 6 months
PTH | Baseline
  For kidney transplant only
1-25 OHD | Baseline
  For kidney transplant only
FGF 23 | Baseline
  For kidney transplant only
calcium | Baseline
  For kidney transplant only
phosphate | Baseline
  For kidney transplant only

CONTACTS AND LOCATIONS:
Overall Officials: Charlene LEVI, Doctor, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Hôpital Femme Mère Enfant, Bron
  - Hopital Edouard Herriot, Lyon
  - CHU Saint Etienne, Saint-Etienne

REFERENCES:
- [Result] De Mul A, Leclerc AS, Ginhoux T, Levi C, Confavreux C, Aurelle M, Portefaix A, Bacchetta J. Changes in bone density and microarchitecture in adolescents undergoing a first kidney transplantation: a prospective study. Eur J Pediatr. 2024 Dec;183(12):5303-5312. doi: 10.1007/s00431-024-05777-z. Epub 2024 Oct 9. PMID 39384649